CLINICAL TRIAL: NCT05299710
Title: Ovarian Tissue Freezing for Fertility Preservation in Pre-Pubertal Children Facing a Fertility Threatening Medical Diagnosis or Treatment Regimen
Brief Title: Ovarian Tissue Cryopreservation in Pre-Pubertal (OTC-Pre Pubertal)
Status: Recruiting | Type: Observational
Sponsor: Erin Rowell (Other)
Collaborators: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Sponsor-Investigator, Erin Rowell, Director of FHPR, Ann & Robert H Lurie Children's Hospital of Chicago
Organization: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Other Study IDs: 2018-1509
Record Dates: First submitted 2020-08-28; First posted 2022-03-29 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Cancers
Keywords: OTC, fertility
MeSH Terms: conditions — Neoplasms; Ornithine Carbamoyltransferase Deficiency Disease | interventions — Laparoscopy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Ovarian Tissue Cryopreservation: Children faced with a fertility threatening diagnosis will be offered ovarian tissue cryopreservation.Pre-surgery assessment will be done while your child is in the hospital or in the pediatric oncology, surgery, or anesthesia clinic as an outpatient. The surgical procedure used to remove your child's ovary is called laparoscopy. It is not required for the treatment of your child's cancer. Laparoscopic surgery is done under general anesthesia (your child will be asleep during the surgery) in the operating room.
  Interventions: Procedure: Laparoscopic surgery

INTERVENTIONS:
Procedure: Laparoscopic surgery — Surgery used to remove your child's ovary tissue is called laparoscopic surgery. Laparoscopic surgery employs a telescope-like instrument called laparoscope. The laparoscope will be put into your child's belly through a small (about half an inch) cut just below the belly button. Two or three other cuts may be made to allow for other instruments to help remove one of the ovaries. The surgeon will then look at both ovaries before the removal of one. Both of your child's ovaries must appear normal and be free of any masses in order to complete the surgery. The surgeon will choose which ovary will be removed at the time of surgery. This type of surgery is likely to last for 30 to 65 minutes.

SUMMARY:
The purpose of this study is to safely remove ovarian tissue in pre-pubertal pediatric patients, who are at risk for infertility from their medical treatment, for freezing for future restoration of fertility and hormone function.

DETAILED DESCRIPTION:
Participants are invited to take part in this study because they will be treated with chemotherapy, radiation and/or surgery that will likely affect the child's ovaries and cause the child to become infertile (unable to become pregnant) in the future.

The ovaries are reproductive glands found only in females. These glands are located in the pelvis (hip area). The ovaries produce eggs and female hormones. During each monthly menstrual cycle, an egg is released from one ovary. This study seeks to find out if removing an ovary in adolescents and children who have reached puberty, and who are about to undergo chemotherapy and/or radiation may preserve, or keep, their ability to have children in the future. The optional ovarian tissue that is removed for research will also be used to study better ways to store the ovarian tissue and to improve of the tissue in the future.

This study has two parts: the removal of the ovarian tissue, and the storage of the ovarian tissue. A process called Ovarian Tissue Cryopreservation will be used to store the removed ovarian tissue. This kind of freezing is a special method that is used to try to prevent the eggs from being damaged, and to keep them frozen for a long time. The frozen tissue will be available to your child to be used at a later time, of your child's choosing.

As a part of the study the investigator is asking participants to donate a 3-4mm biopsy (less than 10% of the ovary) of their ovarian tissue to future research before it is stored for their own use. We also enroll patients in a database study for yearly survey evaluation for long term outcome of ovarian tissue removal and potential restoration.

Ovarian Tissue Cryopreservation involves a surgical procedure where ovarian tissue of post pubertal patients is surgically removed and frozen, with the ultimate goal that their tissue may be used in the future to restore fertility when experimental techniques emerge from the research pipeline. Participation in the study is voluntary.

ELIGIBILITY:
Inclusion Criteria:

* Pre- Pubertal Individual
* Will undergo imminent surgery, chemotherapy or radiation therapy that has implications on future fertility and reproductive hormone potential: any health condition or malignancy that requires removal of all or part of one or both ovaries, whole abdomen or pelvic irradiation ≥10Gy in post-pubertal girls or ≥15Gy in pre-pubertal girls total body irradiation, and alkylating-intensive chemotherapy:
* cyclophosphamide cumulative dose ≥7.5 g/m2
* any treatment regimen containing procarbazine
* busulfan cumulative dose >600 mg/m2
* alkylating chemotherapy conditioning prior to stem cell transplantation combination of any alkylating agent with total body irradiation or whole abdomen or pelvic radiation cranial radiation ≥30 Gy summed alkylating agent dose score ≥3 (Green et al., 2009) cyclophosphamide equivalent dose (CED) ≥ 4,000 mg/m2 (Green et al., 2014)

Exclusion Criteria:

* Patients with no anticipated oncologic therapies
* Post-pubertal individuals
* Pregnant children
* Children with one ovary
* Children deemed high risk for perioperative complications
* Patients unable to provide consent/assent (i.e. significant psychiatric problems/cognitive delay)

Max Age: 11 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — natal females
Study Population: Natal females who have not yet gone through puberty and who face a significant risk of infertility from their medical diagnosis or treatment
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2018-05-29 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2035-01 (Estimated)

PRIMARY OUTCOMES:
Ovarian Tissue Freezing for Fertility Preservation in Pre-Pubertal Children Facing a Fertility Threatening Medical Diagnosis or Treatment Regimen | 3 months
  Most of the surgically removed tissue will be stored for the child's future use. Participants have the option of donating for research purposes a small piece of the ovarian tissue, a small amount of the child's blood and the media used to process the ovarian tissue (which is otherwise discarded, for research which evaluates optimizing ovarian cryopreservation and fertility restoration techniques

SECONDARY OUTCOMES:
Annual follow-up for patients who undergo ovarian tissue cyropreservation | yearly for up to 20 years
  The research study coordinator will contact families by email or telephone once per year and ask a series of questions related to ovarian function, such as beginning puberty and frequency of menstruation.

CONTACTS AND LOCATIONS:
Overall Officials: Erin Rowell, MD, Study Director — Lurie Childrens Hospital
Locations (1):
- Ann & Robert H Lurie Childrens Hospital, Chicago, Illinois, United States

REFERENCES:
- [Background] Armenian SH, Landier W, Hudson MM, Robison LL, Bhatia S; COG Survivorship and Outcomes Committee. Children's Oncology Group's 2013 blueprint for research: survivorship and outcomes. Pediatr Blood Cancer. 2013 Jun;60(6):1063-8. doi: 10.1002/pbc.24422. Epub 2012 Dec 19. PMID 23255494
- [Background] Barton SE, Najita JS, Ginsburg ES, Leisenring WM, Stovall M, Weathers RE, Sklar CA, Robison LL, Diller L. Infertility, infertility treatment, and achievement of pregnancy in female survivors of childhood cancer: a report from the Childhood Cancer Survivor Study cohort. Lancet Oncol. 2013 Aug;14(9):873-81. doi: 10.1016/S1470-2045(13)70251-1. Epub 2013 Jul 13. PMID 23856401
- [Background] Ward E, DeSantis C, Robbins A, Kohler B, Jemal A. Childhood and adolescent cancer statistics, 2014. CA Cancer J Clin. 2014 Mar-Apr;64(2):83-103. doi: 10.3322/caac.21219. Epub 2014 Jan 31. PMID 24488779
- [Background] Martin JR, Kodaman P, Oktay K, Taylor HS. Ovarian cryopreservation with transposition of a contralateral ovary: a combined approach for fertility preservation in women receiving pelvic radiation. Fertil Steril. 2007 Jan;87(1):189.e5-7. doi: 10.1016/j.fertnstert.2006.04.051. Epub 2006 Nov 2. PMID 17084399
- [Background] Paradisi R, Fabbri R, Magnani V, Battaglia C, Venturoli S. A new simple technique of laparoscopic temporary ovarian suspension in addition to ovarian cryopreservation for women prior to posterior pelvic radiation. Gynecol Oncol. 2010 May;117(2):385-6. doi: 10.1016/j.ygyno.2010.01.018. Epub 2010 Feb 13. No abstract available. PMID 20153882
- [Background] Fernbach A, Lockart B, Armus CL, Bashore LM, Levine J, Kroon L, Sylvain G, Rodgers C. Evidence-Based Recommendations for Fertility Preservation Options for Inclusion in Treatment Protocols for Pediatric and Adolescent Patients Diagnosed With Cancer. J Pediatr Oncol Nurs. 2014 Jul;31(4):211-222. doi: 10.1177/1043454214532025. Epub 2014 May 5. PMID 24799444
- [Background] Rowell,EE. Optimal Technique for Laparoscopic Oophorectomy for Ovarian Tissue Cryopreservation in Pediatric Girls In: Woodruff TK GY, ed. Pediatric and Adolescent Oncofertility2017:243-250
- [Background] Practice Committee of American Society for Reproductive Medicine. Fertility preservation in patients undergoing gonadotoxic therapy or gonadectomy: a committee opinion. Fertil Steril. 2013 Nov;100(5):1214-23. doi: 10.1016/j.fertnstert.2013.08.012. Epub 2013 Sep 5. PMID 24011612
- [Background] Hovatta O, Silye R, Krausz T, Abir R, Margara R, Trew G, Lass A, Winston RM. Cryopreservation of human ovarian tissue using dimethylsulphoxide and propanediol-sucrose as cryoprotectants. Hum Reprod. 1996 Jun;11(6):1268-72. doi: 10.1093/oxfordjournals.humrep.a019370. PMID 8671438
- [Background] Filippi F, Meazza C, Paffoni A, Raspagliesi F, Terenziani M, Somigliana E. Egg Freezing in Childhood and Young Adult Cancer Survivors. Pediatrics. 2016 Oct;138(4):e20160291. doi: 10.1542/peds.2016-0291. PMID 27688360
- [Background] Gracia C, Woodruff TK. Oncofertility medical practice : clinical issues and implementation. New York: Springer; 2012
- [Background] Gracia CR, Chang J, Kondapalli L, Prewitt M, Carlson CA, Mattei P, Jeffers S, Ginsberg JP. Ovarian tissue cryopreservation for fertility preservation in cancer patients: successful establishment and feasibility of a multidisciplinary collaboration. J Assist Reprod Genet. 2012 Jun;29(6):495-502. doi: 10.1007/s10815-012-9753-7. Epub 2012 Apr 1. PMID 22466745
- [Background] Duncan FE, Pavone ME, Gunn AH, Badawy S, Gracia C, Ginsberg JP, Lockart B, Gosiengfiao Y, Woodruff TK. Pediatric and Teen Ovarian Tissue Removed for Cryopreservation Contains Follicles Irrespective of Age, Disease Diagnosis, Treatment History, and Specimen Processing Methods. J Adolesc Young Adult Oncol. 2015 Dec;4(4):174-83. doi: 10.1089/jayao.2015.0032. PMID 26697267
- [Background] Jensen AK, Macklon KT, Fedder J, Ernst E, Humaidan P, Andersen CY. 86 successful births and 9 ongoing pregnancies worldwide in women transplanted with frozen-thawed ovarian tissue: focus on birth and perinatal outcome in 40 of these children. J Assist Reprod Genet. 2017 Mar;34(3):325-336. doi: 10.1007/s10815-016-0843-9. Epub 2016 Dec 27. PMID 28028773
- [Background] Demeestere I, Simon P, Dedeken L, Moffa F, Tsepelidis S, Brachet C, Delbaere A, Devreker F, Ferster A. Live birth after autograft of ovarian tissue cryopreserved during childhood. Hum Reprod. 2015 Sep;30(9):2107-9. doi: 10.1093/humrep/dev128. Epub 2015 Jun 9. PMID 26062556
- [Background] Donnelly L. Woman gives birth to baby using ovary frozen in her childhood in 'world first'. The Telegraph 2016
- [Background] Loren AW, Mangu PB, Beck LN, Brennan L, Magdalinski AJ, Partridge AH, Quinn G, Wallace WH, Oktay K; American Society of Clinical Oncology. Fertility preservation for patients with cancer: American Society of Clinical Oncology clinical practice guideline update. J Clin Oncol. 2013 Jul 1;31(19):2500-10. doi: 10.1200/JCO.2013.49.2678. Epub 2013 May 28. PMID 23715580
- [Background] Fallat ME, Hutter J; American Academy of Pediatrics Committee on Bioethics; American Academy of Pediatrics Section on Hematology/Oncology; American Academy of Pediatrics Section on Surgery. Preservation of fertility in pediatric and adolescent patients with cancer. Pediatrics. 2008 May;121(5):e1461-9. doi: 10.1542/peds.2008-0593. PMID 18450888
- [Background] Laronda MM, Jakus AE, Whelan KA, Wertheim JA, Shah RN, Woodruff TK. Initiation of puberty in mice following decellularized ovary transplant. Biomaterials. 2015 May;50:20-9. doi: 10.1016/j.biomaterials.2015.01.051. Epub 2015 Feb 14. PMID 25736492
- [Background] Sorensen SD, Greve T, Wielenga VT, Wallace WH, Andersen CY. Safety considerations for transplanting cryopreserved ovarian tissue to restore fertility in female patients who have recovered from Ewing's sarcoma. Future Oncol. 2014 Feb;10(2):277-83. doi: 10.2217/fon.13.183. PMID 24490613
- [Background] Laronda MM, Duncan FE, Hornick JE, Xu M, Pahnke JE, Whelan KA, Shea LD, Woodruff TK. Alginate encapsulation supports the growth and differentiation of human primordial follicles within ovarian cortical tissue. J Assist Reprod Genet. 2014 Aug;31(8):1013-28. doi: 10.1007/s10815-014-0252-x. Epub 2014 May 21. PMID 24845158
- [Background] Telfer EE, Zelinski MB. Ovarian follicle culture: advances and challenges for human and nonhuman primates. Fertil Steril. 2013 May;99(6):1523-33. doi: 10.1016/j.fertnstert.2013.03.043. PMID 23635350
- [Background] Xiao S, Zhang J, Romero MM, Smith KN, Shea LD, Woodruff TK. In vitro follicle growth supports human oocyte meiotic maturation. Sci Rep. 2015 Nov 27;5:17323. doi: 10.1038/srep17323. PMID 26612176
- [Background] Gosden RG, Telfer E, Faddy MJ, Brook DJ. Ovarian cyclicity and follicular recruitment in unilaterally ovariectomized mice. J Reprod Fertil. 1989 Sep;87(1):257-64. doi: 10.1530/jrf.0.0870257. PMID 2621701
- [Background] Roth JJ, Jones RE. A single ovary of Anolis carolinensis responds more to exogenous gonadotropin if the contralateral ovary is absent. Gen Comp Endocrinol. 1992 Mar;85(3):486-92. doi: 10.1016/0016-6480(92)90093-y. PMID 1577249
- [Background] Khan Z, Gada RP, Tabbaa ZM, Laughlin-Tommaso SK, Jensen JR, Coddington CC 3rd, Stewart EA. Unilateral oophorectomy results in compensatory follicular recruitment in the remaining ovary at time of ovarian stimulation for in vitro fertilization. Fertil Steril. 2014 Mar;101(3):722-7. doi: 10.1016/j.fertnstert.2013.11.019. Epub 2013 Dec 17. PMID 24355047
- [Background] Bjelland EK, Wilkosz P, Tanbo TG, Eskild A. Is unilateral oophorectomy associated with age at menopause? A population study (the HUNT2 Survey). Hum Reprod. 2014 Apr;29(4):835-41. doi: 10.1093/humrep/deu026. Epub 2014 Feb 18. PMID 24549218
- [Background] Wenliang Chen.
- [Background] Gonzalez LP, Pignaton W, Kusano PS, Modolo NS, Braz JR, Braz LG. Anesthesia-related mortality in pediatric patients: a systematic review. Clinics (Sao Paulo). 2012;67(4):381-7. doi: 10.6061/clinics/2012(04)12. PMID 22522764
- [Background] Campo-Engelstein L., Chen D. (2017) Ethical Issues in Pediatric and Adolescent Fertility Preservation. In: Woodruff T., Gosiengfiao Y. (eds) Pediatric and Adolescent Oncofertility. Springer, Cham
- [Background] Nieman CL, Kinahan KE, Yount SE, Rosenbloom SK, Yost KJ, Hahn EA, Volpe T, Dilley KJ, Zoloth L, Woodruff TK. Fertility preservation and adolescent cancer patients: lessons from adult survivors of childhood cancer and their parents. Cancer Treat Res. 2007;138:201-17. doi: 10.1007/978-0-387-72293-1_15. No abstract available. PMID 18080667
- [Background] Gupta AA, Donen RM, Sung L, Boydell KM, Lo KC, Stephens D, Pritchard S, Portwine C, Maloney AM, Lorenzo AJ. Testicular Biopsy for Fertility Preservation in Prepubertal Boys with Cancer: Identifying Preferences for Procedure and Reactions to Disclosure Practices. J Urol. 2016 Jul;196(1):219-24. doi: 10.1016/j.juro.2016.02.2967. Epub 2016 Mar 3. PMID 26947434